CLINICAL TRIAL: NCT00236652
Title: An Open-label, Multi-center, Non-comparative Sinus Puncture Study of 750 mg, Short-course Levofloxacin in the Treatment of Acute Maxillary Sinusitis
Brief Title: A Study Evaluating the Safety and Efficacy of Treating Sinus Infection With Levofloxacin 750 mg for 5 Days.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004678
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Maxillary Sinusitis
Keywords: Maxillary Sinusitis; Infection
MeSH Terms: conditions — Maxillary Sinusitis; Infections | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a once-daily administration of 750 milligrams levofloxacin (an antibiotic) for five days, in treating bacterial sinus infections.

DETAILED DESCRIPTION:
Acute bacterial sinusitis is a common diagnosis for which an antibiotic is prescribed in outpatients. Some types of bacteria that cause sinusitis are resistant to penicillin and certain other classes of antibiotics, but may be treatable with the antibiotic levofloxacin. This will be an open-label, multi-center, non-comparative clinical trial involving outpatients with protocol-defined acute bacterial sinusitis suitable for treatment with oral antibiotics. At the Preliminary Visit, a sinus radiograph will be obtained to confirm the clinical diagnosis of sinusitis, and the Investigator will perform a nasal exam. Sinus puncture and placement of an indwelling sinus catheter into an affected maxillary sinus will be performed on all eligible patients at the first visit. Patients meeting the study criteria will receive 750 milligrams levofloxacin tablets once daily for 5 days. The primary objective is to establish the rate and extent of bacteriological eradication, defined as eradication of pathogens from the maxillary sinus, and to establish the effectiveness and safety of once-daily 750 milligrams levofloxacin for the treatment of acute bacterial sinusitis in adults.

Levofloxacin 750 milligram tablet orally once a day for 5 days

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of acute maxillary sinusitis for 5 to 28 days
* Visible nasal purulence evident on physical examination
* CT scan or standard sinus x-ray (Waters' projections) performed within 5 days prior to the first dose of study drug, showing total sinus opacification or an air-fluid level
* Agree to a maxillary sinus puncture and catheter placement
* If female, using birth control

Exclusion Criteria:

* Chronic sinusitis
* Need for hospitalization or intravenous antibiotics
* History of head, neck, or nasal cancer or surgery
* Previous allergy, serious adverse reaction to, or failed therapy with, levofloxacin or any other member of the quinolone class
* Presence or history of serious complications of sinusitis
* Previous antimicrobial therapy within 7 days of Study Entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-11; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Time to bacteriological eradication, defined as the complete eradication of original strain(s) from the sinus, by the 5th day of levofloxacin treatment.

SECONDARY OUTCOMES:
Efficacy: Clinical response on Day 5 and at the Post-Therapy Visit (Days 12-19); plasma and sinus aspirate concentrations on Days 2-4; levels of inflammatory mediators on Days 0-5. Safety: Adverse events, vital signs, and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Anon JB, Paglia M, Xiang J, Ambrose PG, Jones RN, Kahn JB. Serial sinus aspirate samples during high-dose, short-course levofloxacin treatment of acute maxillary sinusitis. Diagn Microbiol Infect Dis. 2007 Jan;57(1):105-7. doi: 10.1016/j.diagmicrobio.2006.10.019. PMID 17178300
- See also: An Open-Label, Non-Comparative Sinus Puncture Study of 750 MG, Short-Course Levofloxacin in Acute Maxillary Sinusitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=620&filename=CR004678_CSR.pdf